CLINICAL TRIAL: NCT01492816
Title: Enhancement of Connect to Protect® (C2P) to Increase Structural Change and Reduce HIV Risk: Phase IV
Brief Title: Enhancement of Connect to Protect® (C2P)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 105
Record Dates: First submitted 2011-03-22; First posted 2011-12-15 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-05

CONDITIONS: HIV Infection
Keywords: HIV prevention; HIV positive communities
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Group (Experimental): Community members who become engaged in the coalitions and in the broader mobilization effort. A subset of community members.
  Interventions: Behavioral: Community Mobilization

INTERVENTIONS:
Behavioral: Community Mobilization — The proposed study seeks to continue C2P community mobilization efforts that have developed coalitions that plan for and bring about structural changes for purposes of reducing Human Immunodeficiency Virus (HIV) incidence and prevalence among youth in targeted communities at nine sites. Earlier phases of C2P have been outlined in ATN Protocols 016a, 016b, 040/040b. The C2P community mobilization model entails: determining a geographic area and population of focus for the coalitions to prioritize their planning and action (accomplished in an earlier phase of C2P); coalitions establishing a shared vision and mission; development of a strategic plan focused on structural changes to reduce risks associated with HIV; process documentation; and feedback as technical assistance to the coalitions.

SUMMARY:
The proposed study seeks to continue Connect to Protect® (C2P) community mobilization efforts that have developed coalitions that plan for and bring about structural changes for purposes of reducing HIV incidence and prevalence among youth in targeted communities at nine sites.

DETAILED DESCRIPTION:
Earlier phases of C2P have been outlined in ATN Protocols 016a, 016b, 040/040b. The C2P community mobilization model entails: determining a geographic area and population of focus for the coalitions to prioritize their planning and action (accomplished in an earlier phase of C2P); coalitions establishing a shared vision and mission; development of a strategic plan focused on structural changes to reduce risks associated with HIV; process documentation; and feedback as technical assistance to the coalitions. The National Coordinating Center (NCC), operating under the direction of the Protocol Chair, provides guidance, training, technical assistance and feedback to coalitions.

This protocol continues the C2P mobilization effort and includes enhanced strategic planning activities to assist the coalitions in identifying necessary and relevant structural changes. The evaluation of C2P includes both process evaluation (i.e., documentation of coalition actions and achievements of structural changes; and outcome evaluation to qualitatively assess (via Key Informant (KI) interviews) if and how C2P efforts, including completed structural changes, have influenced the risk environment within each community. In addition, local health surveillance data and HIV testing data will be used to evaluate changes in HIV testing patterns and HIV/Sexually Transmitted Infection (STI) morbidity among youth.

ELIGIBILITY:
Inclusion Criteria:

1. The intervention group = Community members who become engaged in the coalitions and in the broader mobilization effort; and
2. The evaluation group = Key Informants within each C2P community who either work or reside within the sectors or systems where structural changes have been accomplished and/or the coalition has focused their strategic planning efforts.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2011-08; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To assess the extent to which C2P activities influence elements of the community that affect HIV-related risk prevention, testing, treatment and linkage to healthcare among youth aged 12-24 years and represent intermediate outcomes for this study. | End of year 5 (study completion)
  Assessment will include evaluation across three primary intermediate outcome areas:
  1. Achievement of SCOs (programs, policies, practices) that target increased levels of HIV-related prevention, testing, and linkage to healthcare.
  2. Increased community capacity and social capital to address HIV-related prevention, testing, and linkage to healthcare.
  3. Increasing levels of sustainability across the HIV continuum of care (CoC) including prevention, testing, and linkage to healthcare activities initiated or influenced by C2P, including programs, policies, and new relationships between people or organizations.

SECONDARY OUTCOMES:
Examine how attributes of the SCOs relate to intermediate outcomes in order to provide guidance and recommendations to policy makers. | End of year 5 (study completion)
  Attributes that will be analyzed include:
  1. Change strategy (e.g., information provision, policy change, relationship formation, program creation).
  2. Sector(s) where change occurs.
  3. Distal vs. proximal causes targeted.
  4. Youth population affected by change (e.g., universal, selected or indicated). In addition, strategies associated with SCO achievement (e.g., creating linkages, honest brokering, strategic partnering, etc.) will be examined for trends and associations.
Assess the trends and associations with strategies used to achieve SCOs (e.g., creating linkages, honest brokering, strategic partnering, etc.) | End of year 5 (study completion)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ellen, MD, Study Chair — Johns Hopkins University Hospital
Locations (9):
- United States (9):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hosp Natinal Med Center, Washington D.C., District of Columbia
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stoger Hospital of Cook County, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: ATN website — http://www.atnonline.org